CLINICAL TRIAL: NCT00853801
Title: Detecting and Managing Metabolic Syndrome and Pre-Diabetes in General Medicine Clinic (Feasibility)
Brief Title: Integrating Lifestyle Therapy for Diabetes Prevention Into Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Leon Fogelfeld MD, Chair, Division of Endocrinology, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MetSyn-PDM
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Pre-Diabetes; Metabolic Syndrome; Type 2 Diabetes
Keywords: Pre-Diabetes; Metabolic Syndrome; Type 2 Diabetes; Diabetes Prevention; Lifestyle Modification; Diet Therapy; Provider Education
MeSH Terms: conditions — Glucose Intolerance; Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Provider/Patient Intervention Arm (Experimental): Lifestyle modification education and counseling for intervention patients. Diagnosis and treatment education and feedback on performance for providers of intervention patients.
  Interventions: Behavioral: Lifestyle intervention and provider feedback
- Provider/Patient Control Arm (No Intervention): Pts will be informed that they have MetSyn and asked to speak with their PCP with any questions.

INTERVENTIONS:
Behavioral: Lifestyle intervention and provider feedback — Patients receive lifestyle education and counseling after each visit with their primary care provider. Lifestyle modification goals are set and progress monitored. Frequency is dependent on frequency of visits with primary care provider which can range from one month to nine months.
  Primary care providers of the intervention patients receive one education session at the commencement of the study covering the diagnosis and treatment of metabolic syndrome and pre-diabetes. Feedback on provider performance as assessed by provider documentation of diagnosis and treatment recommendations compared to patient outcomes is given every six months.
  Arms: Provider/Patient Intervention Arm

SUMMARY:
An educational intervention in the General Medicine Clinic aimed at both primary care providers (PCPs) and their patients with metabolic syndrome/pre-diabetes (MetSyn/PDM). Improving PCPs ability to detect and manage MetSyn/PDM, as measured by the increased incorporation of MetSyn/PDM into PCPs care plan, and increasing patients' awareness of healthy lifestyle behaviors results in positive patient health behaviors and outcomes.

DETAILED DESCRIPTION:
The highest diabetes prevalence in the US is among African Americans (13.3%), American Indians (12.8%), and Mexican Americans (9.5%) with 8.7% of European Americans diagnosed with diabetes. In addition, certain minorities also have much higher rates of diabetes-related complications and death, in some instances by as much as 50% more than the general population, highlighting that the greatest need for preventive measures are amongst ethnic minorities.

The efficacy of lifestyle intervention in reducing the incidence of type 2 diabetes has been established by the Diabetes Prevention Program and other studies. The Cook County Bureau of Health Services, a publicly-funded healthcare system serving a primarily low-income, uninsured, ethnically diverse population in Chicago, IL, currently treats an estimated 40,000 patients annually for type 2 diabetes and estimates that another 85,000 to 100,000 patients are at risk for developing diabetes.

Our primary objective was to test the feasibility of integrating less intensive lifestyle intervention therapy into patient visits with their primary care provider to improve weight loss and decrease the intensity of metabolic syndrome and pre-diabetes risk factors. The site of the study is the General Medicine Clinic, a busy primary care outpatient site treating approximately 12,000 patients/year and 200 patients/day, staffed primarily by medical residents supervised by attending physicians.

ELIGIBILITY:
Inclusion Criteria:

* Has metabolic syndrome as defined by three or more of the five risk factors:

  * elevated blood pressure (BP) above 130 mm Hg systolic and/or 85 mm Hg diastolic or drug therapy for elevated blood pressure
  * elevated waist circumference (WC)above 35" (female) or above 40" (male)
  * reduced high-density lipoprotein (HDL) of below 40 mg/dl (male) or below 50 mg/dl (female) or drug therapy for reduced HDL
  * elevated triglycerides (TG) of 150 mg/dl or above or drug therapy for elevated TG
  * elevated fasting blood glucose (FBG) of 100 mg/dl and above and below 126 mg/dl)or pre-diabetes as defined as elevated FBG.
* Has a primary care provider in the General Medicine Clinic (GMC).

Exclusion Criteria:

* Has been diagnosed with any of the following:

  * diabetes
  * known CAD (MI, CABG, PTCA)
  * congestive Heart Failure NYHA Class III or IV
* Life expectancy less than 2 years
* Non-English speaking patient
* Patient whose physician is a PGY-3 resident, graduating before projected completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-02; Primary Completion 2007-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Patients adopt healthy lifestyle behaviors leading to significant weight loss, thus reducing their risk of diabetes and heart disease | 1.5 years
  Weight loss from baseline
Providers improve their ability to diagnose and treat metabolic syndrome/pre-diabetes. | 1.5 years
  Providers chart MetSyn in Problem List

SECONDARY OUTCOMES:
Improve patient understanding of the metabolic syndrome/pre-diabetes risk parameters and the impact of healthy lifestyle changes on reducing their risk of developing heart disease and diabetes. | 1.5 years
  Patient verbalizes values leading to MetSyn diagnosis
Create a model multidisciplinary team (physician, nurse, dietitian, health educator) to conduct group visits, lifestyle intervention education and follow-up of patients with metabolic syndrome/pre-diabetes. | 1.5 years
  Multidisciplinary team created
Develop a system-wide database of patients with metabolic syndrome/pre-diabetes to target for preventive care. | 1.5 years
  Database developed
Establish physician discussions and documentations encouraging lifestyle changes such as weight loss, healthy dietary changes and exercise. | 1.5 years
  Documentation
Involve nursing staff in waist circumference measurement along with vital signs. | 1.5 years
  Waist measurements documented
Assess changes in insulin resistance using the HOMA-IR index and in vascular inflammation status using C-Reactive protein in the intervention and control groups. | 1.5 years
  HOMA-IR calculated

CONTACTS AND LOCATIONS:
Overall Officials: Leon Fogelfeld, MD, Principal Investigator — Cook County Health
Locations (1):
- John H Stroger Hospital, Chicago, Illinois, United States